CLINICAL TRIAL: NCT01002170
Title: The Impact Factor Analysis of the Therapeutic Drug Monitoring of Oral 2nd Line Antituberculosis Agent, Cycloserine
Brief Title: Pharmacokinetic Study of Patients Who Undergo Cycloserine, a 2nd-line Antituberculosis Medicament
Acronym: CSPK
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Centers for Disease Control, Taiwan (Other Government)
Responsible Party: Ming -Chih Yu, M.D., Chief of Division of Chest Medicine, Taipei Medical University-Wan Fang Hospital
Other Study IDs: TB2NDCSTDMTW
Record Dates: First submitted 2009-07-13; First posted 2009-10-27 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis; Cycloserine; Pharmacokinetics
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In all treatments of tuberculosis, the second-line drugs are usually less effective but have more drug toxicity than the first-line ones. For the multidrug-resistant tuberculosis (MDR-TB) patients, who are resistant to the major first-line anti-tuberculosis drugs such as Rifampin and Isoniazid, the second-line agents, like Cycloserine in this research, are in frequent use. Taking patients' safety into consideration, therapeutic drug monitoring of Cycloserine has been listed as a routine examination during the tuberculosis treatment and established a suggested Cycloserine serum concentration of 20~35 mcg/mL.

While this suggested drug concentration was set up, it isn't suitable to all races in the world. The investigators plan to develop the therapeutic drug monitoring protocols and a suggested treating concentration fitting for Asian (Taiwanese). In addition, through this research, the investigators can also realize that factors causing different pharmacokinetics and the clinical outcomes in different Cycloserine level.

DETAILED DESCRIPTION:
In all treatments of tuberculosis, the second-line drugs are usually less effective but have more drug toxicity than the first-line ones. For the multidrug-resistant tuberculosis (MDR-TB) patients, who are resistant to the major first-line anti-tuberculosis drugs such as Rifampin and Isoniazid, the second-line agents, like Cycloserine in this research, are in frequent use. Taking patients' safety into consideration, therapeutic drug monitoring of Cycloserine has been listed as a routine examination during the tuberculosis treatment and established a suggested Cycloserine serum concentration of 20~35 mcg/mL.

While this suggested drug concentration was set up, it isn't suitable to all races in the world. The investigators plan to develop the therapeutic drug monitoring protocols and a suggested treating concentration fitting for Asian (Taiwanese). In addition, through this research, the investigators can also realize that factors causing different pharmacokinetics and the clinical outcomes in different Cycloserine level.

ELIGIBILITY:
Inclusion Criteria:

* 5 days and more of Cycloserine taking
* Asians

Exclusion Criteria:

* Cancer patients
* AIDS patients
* Combined AIDS-TB patients
* Pregnant subjects
* Anyone whose medical and medication records are unclear

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asia, Taiwan multidrug-resistant tuberculosis (MDR-TB) patients undergo Cycloserine treatment
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Setting up a suggested treating concentration fitting for Asian (Taiwanese) and developing the therapeutic drug monitoring protocols in Taiwan | 2 and 6 hours after dosing

SECONDARY OUTCOMES:
Figuring out that factors causing different pharmacokinetics and the clinical outcomes in different Cycloserine level | 2 and 6 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Yu, M.D., Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan